CLINICAL TRIAL: NCT01973764
Title: Intraventricular Drain Insertion:Comparison of Ultrasound-guided and Landmark-based Puncture of the Ventricular System. A Prospective Randomised Clinical Trial Study.
Brief Title: Intraventricular Drain Insertion: Comparison of Ultrasound-guided and Landmark-based Puncture of the Ventricular System
Acronym: In-Vent
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was stopped due to slow recruitment
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 073/13
Record Dates: First submitted 2013-10-25; First posted 2013-11-01 (Estimated); Last update posted 2019-08-29 (Actual); Status verified 2019-08

CONDITIONS: Hydrocephalus; Intracranial Hypertension
Keywords: Intraoperative ultrasound; Ventricular System; Puncture; Ventricular catheter; Ventriculostomy; Hydrocephalus; Excessive accumulation of cerebrospinal fluids within the cranium. Often associated with dilatation of cerebral ventricles; Intracranial Hypertension; increased pressure within the cranial vault. This may result from several conditions, including hydrocephalus, brain edema.
MeSH Terms: conditions — Hydrocephalus; Intracranial Hypertension; Brain Edema

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ultrasound guided arm (Other)
  Interventions: Procedure: Ultrasound guided ventricular drain insertion
- Landmark-based arm (Other)
  Interventions: Procedure: landmark-based ventricular drain insertion

INTERVENTIONS:
Procedure: Ultrasound guided ventricular drain insertion — Ventricular puncture and insertion of the intraventricular catheter is performed under ultrasound guidance.
  Arms: Ultrasound guided arm
Procedure: landmark-based ventricular drain insertion — Ventricular puncture and insertion of the intraventricular catheter is performed without any guiding devices and is based on anatomical landmarks.
  Arms: Landmark-based arm

SUMMARY:
Puncture of the ventricular system is one of the most frequently performed neurosurgical interventions. This procedure is commonly performed in order to treat and/or measure pathologically elevated intracranial pressure.Therefore a safe and fast surgical procedure is needed. Currently the "landmark-based" placement of intraventricular catheters is the gold standard. However it is known that more than 60% of the catheters are not accurately placed in accordance with "landmark-based" procedures. When the catheter is not placed accurately multiple punctures may be required. In this study, the investigators aim to investigate prospectively whether ultrasound guidance leads to a lower number of incorrect catheter placements, and whether this guidance consequently decreases the number of punctures.

DETAILED DESCRIPTION:
Background

Puncture of the ventricular system is one of the most frequently performed neurosurgical interventions. This procedure is performed in order to treat and/or measure pathologically elevated intracranial pressure. Therefore a safe and fast surgical procedure is needed. Currently the "landmark-based" placement of intraventricular catheters is the gold standard. Nonetheless it is known that more than 60% of the catheters are not placed accurately performing "landmark-based" procedures. When the catheter is not placed accurately multiple punctures may has to be done.

Puncture of the ventricular system is one of the most frequently performed neurosurgical interventions. This procedure is commonly performed in order to treat and/or measure pathologically elevated intracranial pressure. Therefore a safe and fast surgical procedure is needed.Currently the "landmark-based" placement of intraventricular catheters is the gold standard. Nonetheless it is known that more than 60% of the catheters are not placed accurately performing "landmark-based" procedures. When the catheter is not placed accurately multiple punctures may be required. Incorrectly placed intraventricular catheters may lead to undesirable side effects like catheter dysfunction,in which case a correction of the catheter position or a even a new puncture will be required. These corrections increase the risk of intracerebral hemorrhages, infections or secondary brain injuries. In this study, the investigators will prospectively investigate whether ultrasound guidance increases the number of well-placed ventricular catheters and reduces the number of undesirable side effects. In this study the correct catheter position is defined when the catheter tip is located in the lateral ventricle (ipsilateral to the burrhole) anterior of the foramen of Monro. Catheter tip position will be assessed by cranial computer tomography after the operation. The CT scans will be evaluated by an independent expert rater, blinded for the procedure type. These incorrectly placed intraventricular catheters may lead to undesirable side effects, like catheter dysfunction wherefore a correction of the catheter position or a even a new puncture has to be done. These corrections increase the risk of intracerebral hemorrhages, infections or secondary brain damages.

In this study, the investigators will prospectively investigate if ultrasound guidance may raise the number of well placed ventricular catheters and may reduce the number of undesirable side effects. In this study the correct catheter position is defined when the catheter tip is located in the ipsilateral lateral ventricle (to the burrhole) anterior of the foramen of monroi and will be assessed by cranial computer tomography after operation. The CT Scans will be evaluated by an independent expert rater, blinded for the procedure type.

Objective

Aim of the study is to investigate whether ultrasound guidance of ventricular catheter placement leads to a lower number of incorrectly placed catheters and lower number of punctures compared to the landmark-based procedure.

Methods

This study is a prospective randomized controlled clinical trial. A total of 90 patients will be included in the study and randomized in two groups with 45 patients each (ultrasound-guided group and landmark-based group). The position of the ventricular catheter will be assessed using cranial computer tomography (CCT). The CT Scans will be evaluated by two independent expert raters, blinded for the procedure type.

ELIGIBILITY:
Inclusion Criteria:

* Age >/= 18 years
* Intraventricular catheter insertion or/and intraventricular pressure measurement indicated
* Written informed consent

Exclusion Criteria

* Age < 18 years
* previous ventricular punction < 4 weeks
* bedside puncture indicated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2013-11; Primary Completion 2019-05 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
The correct ventricular catheter position (on post op CT) after single ventricular puncture. | 48 h after initial operation

SECONDARY OUTCOMES:
Number of catheter changes | at hospital discharge, expected to be after 10 days
Number of infections | at hospital discharge, expected to be after 10 days
Number of days in clinic | at hospital discharge, expected to be after 10 days
Number of ventricular punctures | "at the end of the operation, expected to be after 1 hour"
Number of patients with intracerebral hemorrhage | 24 h after initial operation

CONTACTS AND LOCATIONS:
Overall Officials: Jürgen Beck, MD, Principal Investigator — Dep. of Neurosurgery, University Hospital Bern; Andreas Raabe, MD, Study Director — Dep. of Neurosurgery, University Hospital
Locations (1):
- Dep. of Neurosurgery, Bern University Hospital, Bern, Switzerland

REFERENCES:
- [Result] Toma AK, Camp S, Watkins LD, Grieve J, Kitchen ND. External ventricular drain insertion accuracy: is there a need for change in practice? Neurosurgery. 2009 Dec;65(6):1197-200; discussion 1200-1. doi: 10.1227/01.NEU.0000356973.39913.0B. PMID 19934980
- [Result] Sekhar LN, Moossy J, Guthkelch AN. Malfunctioning ventriculoperitoneal shunts. Clinical and pathological features. J Neurosurg. 1982 Mar;56(3):411-6. doi: 10.3171/jns.1982.56.3.0411. PMID 7057239
- [Result] Pang D, Grabb PA. Accurate placement of coronal ventricular catheter using stereotactic coordinate-guided free-hand passage. Technical note. J Neurosurg. 1994 Apr;80(4):750-5. doi: 10.3171/jns.1994.80.4.0750. PMID 8151359
- [Result] Huyette DR, Turnbow BJ, Kaufman C, Vaslow DF, Whiting BB, Oh MY. Accuracy of the freehand pass technique for ventriculostomy catheter placement: retrospective assessment using computed tomography scans. J Neurosurg. 2008 Jan;108(1):88-91. doi: 10.3171/JNS/2008/108/01/0088. PMID 18173315
- [Result] Wilson TJ, Stetler WR Jr, Al-Holou WN, Sullivan SE. Comparison of the accuracy of ventricular catheter placement using freehand placement, ultrasonic guidance, and stereotactic neuronavigation. J Neurosurg. 2013 Jul;119(1):66-70. doi: 10.3171/2012.11.JNS111384. Epub 2013 Jan 18. PMID 23330995
- [Result] Strowitzki M, Moringlane JR, Steudel W. Ultrasound-based navigation during intracranial burr hole procedures: experience in a series of 100 cases. Surg Neurol. 2000 Aug;54(2):134-44. doi: 10.1016/s0090-3019(00)00267-6. PMID 11077095
- [Result] Maniker AH, Vaynman AY, Karimi RJ, Sabit AO, Holland B. Hemorrhagic complications of external ventricular drainage. Neurosurgery. 2006 Oct;59(4 Suppl 2):ONS419-24; discussion ONS424-5. doi: 10.1227/01.NEU.0000222817.99752.E6. PMID 17041512